CLINICAL TRIAL: NCT05601622
Title: Assessment of Predictive Power for Fluid Responsiveness of Rainbow Pleth Variability Index in Children
Brief Title: RPVI for Fluid Responsiveness in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2209-123-1363
Record Dates: First submitted 2022-10-20; First posted 2022-11-01 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Fluid Responsiveness
Keywords: Fluid responsiveness; pleth variability index
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Fluid loading, Stroke volume index measurement via transthoracic echocardiography, measurement of pleth variability index and Rainbow pleth variability index, change of tidal volume under mechanical ventilation
  Interventions: Procedure: Fluid loading; Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: PVI, RPVI; Procedure: Tidal volume change

INTERVENTIONS:
Procedure: Fluid loading — Intravenous administration of 10ml/kg of crystalloids over 10 minutes
Diagnostic Test: Transthoracic echocardiography — Transthoracic echocardiographic measurement of stroke volume index
Diagnostic Test: PVI, RPVI — Continuous measurement of pleth variability index and Rainbow pleth variability index
Procedure: Tidal volume change — Changing tidal volume for mechanical ventilation as 6, 8, 10 ml/kg

SUMMARY:
The purpose of this study is to validate Rainbow pleth variability index for prediction of fluid responsiveness in children.

DETAILED DESCRIPTION:
Children undergoing surgery under general anesthesia will be enrolled. After anesthetic induction, they will be assessed via transthoracic echocardiography for measurement of the patient's stroke volume index (SVI). Also, pleth variability index and Rainbow pleth variability index will be measured under mechanical ventilation with tidal volume of 6, 8, 10 ml/kg.

To exert fluid loading, 10ml/kg of crystalloid solution will be administered intravenously over 10 minutes. After fluid loading, the SVI will be measured again and fluid responsiveness will be determined according to increment ratio of the SVI.

According to the determined fluid responsiveness, predictive power of pleth variability index and Rainbow pleth variability index for fluid responsiveness will be assessed by building a receiver-operating characteristics curve.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing neurosurgery under general anesthesia

Exclusion Criteria:

* Presence of any cardiovascular disease
* Presence of any pulmonary disease
* Decline of enrollment from any of the patient's parents

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
AUC of ROC curve | From start of anesthesia to end of anesthesia, Less than 24 hours
  Area under the curve of the receiver-operating characteristics curve of pleth variability index and Rainbow pleth variability index for prediction of fluid responsiveness

SECONDARY OUTCOMES:
Appearance of abnormal heart rhythm | From start of anesthesia to end of study, Less than 24 hours
  Electrocardiogram during the study for monitoring whether tachycardia, bradycardia, or arrhythmia appears. Heart rate will be compared between patients who were fluid responsive and who were not responsive.
IBP | From start of anesthesia to end of study, Less than 24 hours
  Invasive blood pressure during the study, including systolic, diastolic, mean blood pressure for monitoring whether hypertension or hypotension appears. Mean blood pressure will be compared between patients who were fluid responsive and who were not responsive.
SpO2 | From start of anesthesia to end of study, Less than 24 hours
  Pulse oximetry during the study for monitoring whether hypoxia appears.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan H, Cannesson M, Chandler JR, Ansermino JM. Predicting fluid responsiveness in children: a systematic review. Anesth Analg. 2013 Dec;117(6):1380-92. doi: 10.1213/ANE.0b013e3182a9557e. PMID 24257389
- [Background] Han YY, Carcillo JA, Dragotta MA, Bills DM, Watson RS, Westerman ME, Orr RA. Early reversal of pediatric-neonatal septic shock by community physicians is associated with improved outcome. Pediatrics. 2003 Oct;112(4):793-9. doi: 10.1542/peds.112.4.793. PMID 14523168
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169